CLINICAL TRIAL: NCT04908553
Title: Safety and Dose Exploration of Remimazolam Tosilate for Injection for Induction and Maintenance of General Anesthesia Intubation for Elective Short-term Surgery in Adults: a Multi-center, Randomized, Double-blind Clinical Study
Brief Title: Study on the Safety and Effectiveness of Remimazolam Tosilate for Injection for Short-term Elective Surgery in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ailin Luo, Principal Investigator, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021S027
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hypotension During Surgery
MeSH Terms: interventions — Injections; Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Other): Remimazolam Tosilate for Injection 0.1mg/kg at induction
  Interventions: Drug: Remimazolam Tosilate for Injection 0.1mg/kg
- medium dose group (Other): Remimazolam Tosilate for Injection 0.15mg/kg at induction
  Interventions: Drug: Remimazolam Tosilate for Injection 0.15mg/kg
- high dose group (Other): Remimazolam Tosilate for Injection 0.2mg/kg at induction
  Interventions: Drug: Remimazolam Tosilate for Injection 0.2mg/kg

INTERVENTIONS:
Drug: Remimazolam Tosilate for Injection 0.1mg/kg — Remimazolam Tosilate for Injection 0.1mg/kg at induction
  Other Names: low dose group
  Arms: low dose group
Drug: Remimazolam Tosilate for Injection 0.15mg/kg — Remimazolam Tosilate for Injection 0.15mg/kg at induction
  Other Names: medium dose group
  Arms: medium dose group
Drug: Remimazolam Tosilate for Injection 0.2mg/kg — Remimazolam Tosilate for Injection 0.2mg/kg at induction
  Other Names: high dose group
  Arms: high dose group

SUMMARY:
Research objective: To explore the safety and dose exploration of Remimazolam Tosilate for Injection for induction and maintenance of general anesthesia in elective short-term surgery in adults.

Main research indicators:(1)Success rate of sedation during induction and maintenance of general anesthesia with remazolam tosylate;(2)The incidence and severity of hypotension in the induction and maintenance phases Study design: Multi-center, randomized, double-blind clinical study. Subject population: patients undergoing elective short-term surgery. Research data collection period: The subject signs the consent form until discharge or death in the hospital or withdrawal from the research.

Number of research centers/sample size: It is planned to enroll 600 patients from 11 hospitals.

Research process: The researchers will include patients who meet the enrollment criteria and agree to participate in the investigation of the support laryngoscope surgery and minor head and neck surgery patients from the elective surgery patients.

DETAILED DESCRIPTION:
The data collected in this study is recorded by the researcher in the eCRF, including:

1. Data to be collected during the screening period and before the operation: the basic characteristics of the patient and demographic data;
2. Data to be recorded during and/or postoperatively: main research indicators, secondary indicators and other indicators.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ-Ⅲ grade;
2. age 18-65 years old;
3. gender is not limited;
4. planned elective support laryngoscope surgery (glottic polypectomy under support laryngoscope, epiglottic cyst excision under support laryngoscope, benign laryngeal under support laryngoscope Lesion resection), endoscopic septoplasty, endoscopic tympanoplasty, endoscopic middle ear tube insertion, nasopharyngoplasty, head and neck benign mass resection for general anesthesia intubation patients;
5. operation time No more than 90min.

Exclusion Criteria:

- Emergency surgery;

1. abnormal renal function (urea nitrogen ≥1.5×ULN, blood creatinine greater than the upper limit of normal);
2. abnormal liver function;
3. hypovolemia, shock or coma;
4. suffering from mental illness and long-term use of psychotropic drugs;
5. cognition Dysfunction;
6. those who are allergic to or contraindicated to benzodiazepines and their drug components; pregnant or lactating female patients;
7. have a history of drug dependence;
8. have used other sedatives in the past week;
9. have been a subject within the past 3 months Participated in drug clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension during the anesthesia | during the anesthesia procedure
  The systolic blood pressure during the anesthesia is ≤ 90 mmHg, or a reduction of >20% from the baseline period, or the average blood pressure is <65 mmHg
The rate of Successful sedation during the anesthesia | during the anesthesia procedure
  Successful sedation during the anesthesia is defined as: 1) successful induction of anesthesia without anesthesia remedial measures during the induction period; 2) no recovery during the anesthesia maintenance period, no unexpected physical activity, and no remedial measures during the maintenance period anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No